CLINICAL TRIAL: NCT06669663
Title: Hypoxia Driven Metabolic Response in Oesophagogastric Adenocarcinoma
Acronym: HYDRA
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 324771; MR/Z504142/1 (Other Grant/Funding Number: Medical Research Council); 23/PR/0723 (Registry Identifier: Human Research Authority (HRA) Research Ethics Council (REC))
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: OESOPHAGO-GASTRIC CARCINOMA
Keywords: voc; hypoxia; pimonidazole; oesophago-gastric carcinoma; volatile organic compounds; breath test
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour Tissue Pimonidazole Labelled Tumour Tissue Breath Urine Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pimonidazole Group: Will receive Pimonidazole (as a non-CTIMP) to enable hypoxic tumour stratification
  Interventions: Drug: Pimonidazole hydrochloride (Hypoxyprobe™-1)
- Biosampling Group: Participants will undergo blood, urine and breath sampling on their morning of their surgery on their OG tumour. Intra-operatively, tumour samples will be taken.

INTERVENTIONS:
Drug: Pimonidazole hydrochloride (Hypoxyprobe™-1) — Participants will receive Pimonidazole (non-CTIMP) prior to their surgery for OG cancer and then undergo intra-operative sampling.
  Groups: Pimonidazole Group

SUMMARY:
Oesophagogastric Cancer and Hypoxia:

Oesophagogastric cancer is a significant global burden, with 1.7 million new cases per year. It is well known that survival from oesophagogastric cancer is poor. Five-year survival for these cancers in the UK remains between 15-20%, which is amongst the lowest in Europe. The reason for this poor survival is multifactorial, with late diagnosis and treatment-resistant hypoxic tumours both significantly contributing to this high mortality.

Tumour hypoxia occurs when rapidly growing malignancies outstrip oxygen (and nutrient) supply. These hypoxic conditions trigger adaptive metabolic and genomic mutations within the cancer. Clinically, these mutations lead to cancers which are highly aggressive and treatment resistant. Therefore, patients with oesophagogastric cancers displaying high degrees of hypoxia have a considerably poorer prognosis. Reassuringly, there are emerging treatment options available. The adaptive pathways triggered by hypoxia offer unique opportunities for personalized and targeted oncological therapies to improve clinical outcomes in this patient cohort. However, for these therapies to be effective, it is vital patients with hypoxic tumours can be identified.

There are currently no established methods for identifying hypoxic tumours in oesophagogastric cancer patients. Whilst biomarker candidates have been identified, these require invasive biopsies and are limited in terms of repeatability, and therefore clinical applicability. There is hope in developing non-invasive hypoxic imaging, however considerable validation work is required prior to their clinical introduction for oesophagogastric patients.

Volatile Organic Compounds and Breath:

The Hanna Group at Imperial College London has developed a non-invasive breath test for the diagnosis of oesophagogastric adenocarcinoma through the detection of exhaled Volatile Organic Compounds (VOCs). This was validated in a multi-centre NIHR-funded clinical study that demonstrated 80% sensitivity and 81% specificity. In parallel with this work, the exhalation kinetics and molecular drivers of VOCs in oesophagogastric adenocarcinoma have also been investigated. It has been understood that the VOCs that can be detected in blood, breath, urine, and saliva are a representation of the metabolic and microbiotic changes that occur in the tumour and its microenvironment.

Rationale for Study:

There is a clear unmet need for a dynamic non-invasive test to identify patients suffering with hypoxic oesophagogastric tumours. By adapting the breath test model, it is believed that patients with hypoxic tumours can be effectively detected. This creates the opportunity to offer targeted oncological therapies for these patients. Furthermore, the reproducibility and patient acceptability make a breath test an ideal testing method for dynamic hypoxia monitoring .

Promising work within the Hanna Group has already demonstrated the potential viability of a 'hypoxia breath test'. Early cell culture experiments and pilot studies have demonstrated hypoxic tumours release discriminatory VOCs which could be leveraged as hypoxic biomarkers.

HYDRA Study

The HYDRA study is a single-centre observational study at Imperial College London with the aim of devising a non-invasive breath test for OG tumour hypoxia. The study contains two arms: the Pimonidazole and Biosampling arm.

In the Pimonidazole arm, 20 participants (10 oesophageal and 10 gastric cancer) will be given Pimonidazole (Hypoxyprobe Inc.), a hypoxia-labelling agent, prior to their surgery for oesophagogastric cancer. Hypoxia-stratified tissue will be sampled intraoperatively and analysed using spatial transcriptomics and spatial metabolomic techniques. This will allow the creation of an OG-hypoxic gene signature.

The Biosampling arm will recruit 100 patients undergoing OG cancer surgery. Participants will undergo breath sampling and intra-operative tumour sampling. Using the hypoxic gene signature generated in the Pimonidazole arm, transcriptomic analysis of tumour samples will allow patient categorisation into hypoxia-high and hypoxia-low subgroups. This will enable our group to devise a hypoxic OG breath test, separating patients with hypoxia-high and hypoxia-low tumours.

ELIGIBILITY:
Inclusion Criteria:

* Male and females aged 18-90 years.
* Patients with biopsy proven oesophageal or gastric adenocarcinoma who are undergoing either surgical resection or staging laparoscopy.

Exclusion Criteria:

* Non-adenocarcinoma cancer (e.g. oesophageal squamous cell carcinoma)
* Antibiotic therapy within the last 8 weeks
* Previous oesophageal and gastric resection
* Allergy to pimonidazole
* Unable or unwilling to provide informed written consent
* Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oesophago-gastric patients undergoing surgery on their cancer
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Hypoxic Gene Signature | 5 years
  Spatial transcriptomic, lipidomic and pathway analysis on pimonidazole-labelled tissue will allow the identification of a OAC hypoxic gene signature.
Volatile Organic Compounds Breath Signature | 5 years
  Bulk RNAseq will be performed on tumour samples from Biosampling participants. Participants will then be classified by their hypoxic score using the previously derived hypoxic gene signature. Distinguishing Volatile Organic Compounds (VOCs) detected in exhaled breath, using GC-MS, between these two groups will generate an OAC hypoxic breath profile.

CONTACTS AND LOCATIONS:
Overall Officials: George Hanna, Principal Investigator — Imperial College London; Henry Robb, MBChB BSc (Hons) MSc MRCS, Study Director — Imperial College London; Bibek Das, MBChB, Study Chair — Imperial College London
Locations (1):
- Imperial College NHS Healthcare Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No